CLINICAL TRIAL: NCT02126358
Title: A Multicenter, Randomized, Placebo-controlled, Double-blind, Phase III Trial to Evaluate the Efficacy and Safety of the Fix-dose Combination Therapy With Gemigliptin 50mg and Rosuvastatin 20mg With Type 2 Diabetes and Dyslipidemia
Brief Title: Gemigliptin-Rosuvastatin Fix-dose Combination Phase 3(BALANCE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LG-GSCL002
Record Dates: First submitted 2014-03-04; First posted 2014-04-30 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gemigliptin (Placebo Comparator): only Gemiglitpin (Gemiglitpin/Rosuvastatin FDC:Placebo , Rosuvastatin :Placebo)
  Interventions: Drug: Gemigliptin and/or Rosuvastatin
- Rosuvastatin (Placebo Comparator): only Rosuvastatin (Gemiglitpin/Rosuvastatin FDC:Placebo , gemigliptin :Placebo)
  Interventions: Drug: Gemigliptin and/or Rosuvastatin
- FDC (Experimental): Gemigliptin & Rosuvastatin (Gemiglitpin only:Placebo ,Rosuvastatin only:Placebo)
  Interventions: Drug: Gemigliptin and/or Rosuvastatin

INTERVENTIONS:
Drug: Gemigliptin and/or Rosuvastatin

SUMMARY:
To evaluate the efficacy and safety of the fix-dose combination therapy with Gemigliptin 50mg and Rosuvastatin 20mg with type 2 diabetes and dyslipidemia

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus with Dyslipidemia
* Adults who are at least 19 years old

Exclusion Criteria:

* Patients with type 1 diabetes, diabetic ketoacidosis, diabetic coma and pre-coma
* Patients with gestational diabetes or secondary diabetes
* Patients with NYHA Class III, IV congestive heart failure or arrhythmias requiring treatment
* Patients with thyroid gland dysfunction deviating from the normal TSH range
* Patients with pituitary insufficiency or adrenal insufficiency

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
HbA1c change | Baseline(Day 0) to Treatment (last visit, w24)
LDL-C change rate | Baseline(Day 0) to Treatment (last visit, w24)

SECONDARY OUTCOMES:
HbA1c | Baseline(Day 0) to Treatment (last visit, w24)
  (Gemigliptin/Rosuvastatin FDC vs. Gemigliptin)
LDL-C change rate | Baseline(Day 0) to Treatment (last visit, w24)
  (Gemigliptin/Rosuvastatin FDC vs. Rosuvastatin)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, South Korea